CLINICAL TRIAL: NCT03566186
Title: Effects of Phototherapy Associated With Sprint and Squat Training on Cardiac Autonomic Modulation: Randomized, Placebo-controlled Trial
Brief Title: Effects of Phototherapy Associated With Sprint and Squat Training on Cardiac Autonomic Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, PhD - Clinical Professor, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: U1111-1214-0497
Record Dates: First submitted 2018-05-28; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Phototherapy; Autonomic Nervous System; Training
Keywords: Photobiomodulation; Autonomic nervous system; Heart rate variability; Recovery of function; Super-pulsed laser; Led light
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active phototherapy group (Experimental): (n=12) Phase 2 training + active phototherapy Dosage applied was 30J per site (180J per muscle) to six sites on the quadriceps The MR4 LaserShower 50 4D emitter (MultiRadiance Medical, USA). The optical power was calibrated before irradiationin each participant using a Thorlabs thermal power meter(Model S322C, Thorlabs, Newton, NJ, USA).
  Interventions: Other: Phototherapy
- Placebo group (Placebo Comparator): (n=14) Phase 2 training + placebo phototherapy group
  Interventions: Other: Placebo
- non-treatment control group (Other): (n=13) Phase 2 training + control group
  Interventions: Other: Passive recovery

INTERVENTIONS:
Other: Phototherapy — Photobiomodulation or photobiostimulation, this technique is the application of monochromatic light that can influence cellular activity through inhibition or stimulation of chemical and biological functions.
  Arms: Active phototherapy group
Other: Placebo — The same procedures as in the active phototherapy group was applied to the placebo group; however, the emitter was disabled. The device was emit the same sounds regardless of the programmed mode (active phototherapy).
  Arms: Placebo group
Other: Passive recovery — Participants was remain sat for passive recovery supervised by an independent therapist during the period when the other groups are received recovery strategies.
  Arms: non-treatment control group

SUMMARY:
Recent studies have shown positive results in the application of phototherapy for the improvement of performance and acceleration of the healing process of the body homeostasis. Among the methods used to assess the recovery post-exercise has cardiac autonomic modulation assessed by heart rate variability (HRV), a tool widely used in sports to evaluate medium global behavior of the autonomic nervous system. Objective: analyze and compare the effect of a special protocol of phototherapy using different light sources interacting with a combined training with an autonomic modulation of heart rate in different moments (baseline; tracking daily; recovery post-exercise and after training). Method: 45 male participants will be allocated from a stratified randomization into three groups: control (n=15), placebo (n=15) and group special protocol of phototherapy (n=15). Participants will perform a combined training of sprints and squats twice a week for twelve weeks divided into two phases. The application of phototherapy and placebo was administered in phase 2, after sprints and just before the squat. The phototherapy was used combine different light sources and wavelength (red and infrared). Was analyze HRV in five moments: baseline; traking daily; week target of phase I and II; after training. The weeks target consist of training sessions with greater energy expenditure (largest intensity). The sphericity of the data was tested by Mauchly test. In case of violation of the sphericity assumption, the correction of Greenhouse-Geisser was performed. The data was analyzed using analysis of variance for repeated measures (Bonferroni post-test), which provide information on the effects of time, group and interaction. All statistical analyzes assume the significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient (self-report);
* Male gender;

Exclusion Criteria:

* History of cancer;
* Smokers or alcoholics;
* Use drugs that influenced cardiac autonomic activity;
* Cardiovascular, metabolic or endocrine diseases;
* Occurrence of musculoskeletal injury during the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-03 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Effects of phototherapy on adaptation and change of cardiac Autonomic modulation. | Baseline (captation of hear rate variability for 20 minutes) before 6 weeks (captation of hear rate variability for 20 minutes) and before 12 weeks (captation of hear rate variability for 20 minutes)
  Analyzed and compare the effects of phototherapy with different light sources and wavelengths applied during training combined at heart rate variability

SECONDARY OUTCOMES:
Effects of phototherapy on recovery of cardiac Autonomic modulation. | During training sessions with higher energetic spending leaving for the last two weeks, composed of higher intensity - (captation of hear rate variability for 1 hour on phase 1 and phase 2).
  Compare the effects of phototherapy with placebo group and control group at recovery after exercise of heart rate variability.
Effects of phototherapy on tracking daily of cardiac autonomic modulation. | daily, after exercise and before exercise (captation of hear rate variability for 7 minutes)
  Analyze and compare the change in the indices of heart rate variability in tracking daily after combined training of sprints and squats

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil